CLINICAL TRIAL: NCT04211181
Title: Effect on Thromboprophylaxis Among Hospitalized Patients Using a System-wide Multifaceted Quality Improvement Intervention: Rationale and Design for a Multicenter Cluster Randomized Clinical Trial in China
Brief Title: CHIPs-VTE Study in Hospitalized Patients to Prevent Hospital-Acquired Venous Thromboembolism
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Zhenguo Zhai,MD,PhD, Principal investigator, China-Japan Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CHIPs-VTE in inpatient
Record Dates: First submitted 2019-12-08; First posted 2019-12-26 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Venous Thromboembolic Disease; Pulmonary Embolism; Venous Thromboembolism; Deep Venous Thrombosis; Quality Improvement
Keywords: Quality improvement; Venous Thromboembolism; Hospital Associated-VTE
MeSH Terms: conditions — Pulmonary Embolism; Venous Thromboembolism; Venous Thrombosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The multifaceted QI interventions (Experimental): Hospitals randomized into experimental group will implement follow interventions including：the distribution of the guideline and pathway, a computer alert(computer-based clinical decision support system and computerized reminders),audit and feedback.
  Interventions: Other: The multifaceted interventions
- Routine VTE prophylaxis in local clinical practice (Active Comparator): Patients in the routine VTE prophylaxis(control) group will receive routine VTE prophylaxis according to current guidelines and clinical practices.
  Interventions: Other: Routine VTE prophylaxis

INTERVENTIONS:
Other: The multifaceted interventions — 1. An evidence-based clinical guideline and pathway in hospital.
  2. A series Written care protocols for the implementation of performance measures.
  3. A newly developed mobile application (mini-program) will be employed to facilitate venous thromboembolism (VTE) risk assessment and prophylaxis. Patients will scan a QR code to enroll in the program and be linked with their physician. Through the application, patients will complete standardized self-assessments of VTE risk, and physicians will receive periodic reminders indicating whether the assessment and prophylaxis orders have been completed.The application also provides educational modules and targeted messages for both patients and physicians, and enables interactive communication.
  4. A quality-control team will receive weekly feedback reports to verify whether all enrolled patients underwent appropriate prophylaxis.
  Arms: The multifaceted QI interventions
Other: Routine VTE prophylaxis — Patients randomized to the Routine VTE prophylaxis (Control) group will receive routine VTE prophylaxis according to current guidelines and clinical practices
  Arms: Routine VTE prophylaxis in local clinical practice

SUMMARY:
Although pharmacologic and mechanical methods to prevent VTE are safe, effective, cost-effective, and advocated by authoritative guidelines,many studies continue to demonstrate that these preventive methods are significantly underutilized, especially in China.A number of quality improvements (QI) program have been established in several countries or hospitals.However,no exit effective protocol has been demonstrated well enough or adequate to drive breakthrough levels of improvement. A reliable and practical QI that can support hospitals or physicians in China is warranted.To evaluate the multifaceted quality improvement intervention effect in clinical setting, we will conduct a cluster-randomized clinical trial among China PUlmonary Thromboembolism REgistry Study (CURES) group, aiming to test whether it's applicable to real-world practice in China.

A multicenter, two-arms, open-label clinical trial has been designed to determine whether the system-wide multifaceted intervention could increase the rate of at-risk participants who received prophylaxis (RP) and decrease the incidence of any hospital-associated VTE in 90 days during and after hospital admission. .Selected hospital will be regarded as a cluster and randomized into interventional or control group.In interventional group, eligible hospitalized patients will receive a variety of the multifaceted quality improvement(QI) interventions since admitted in hospital.In control group, patients will receive no more than common recommended care or an existing policy.The primary outcomes are the proportion of appropriate prophylaxis in hospitalized patients and the incidence of HA-VTE in 90 days after hospital admission.

DETAILED DESCRIPTION:
Hospitals nationwide which have willingness to participate this study in CURES group will be selected. Each selected hospital will be regarded as a cluster and randomized into interventional or control group.

During the study period, eligible patients enrolled in hospitals assigned to interventional group will receive a variety of the multifaceted quality improvement(QI) interventions, including mandatory risk assessment, a computer alert(computer-based clinical decision support system and computerized reminders), strengthened education, and audit. Patients in hospitals assigned to control group will receive common recommended care only, or an existing policy.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥14 years
2. Have an expected hospital stay ≥72 hours for medical and/or surgical treatment
3. Written informed consent

Exclusion Criteria:

1. Inability to be followed-up at until 3 months after randomization
2. Have participated in similar trials or are undergoing other clinical trials
3. Refuse or are unable to give informed consent
4. VTE identified on CTPA or lower extremity vein ultrasound at or any time before enrollment
5. Requiring a full dose of anticoagulant treatment (e.g., recent VTE, atrial fibrillation).

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5800 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of appropriate prophylaxis rate during hospitalization | 90 days after hospital admission
  The proportion of appropriate prophylaxis is defined as the number of appropriate prophylaxis among the patients at risk of VTE and without corresponding contraindications.
The proportion of participants who developed the VTE(all, symptomatic, asymptomatic VTE) | 90 days after hospital admission
  The incidence of HA-VTE is defined as the proportion of participants who developed the VTE(all, symptomatic, asymptomatic VTE)

SECONDARY OUTCOMES:
All-cause mortality | 90 days after hospital admission
  Proportion of participants who was dead(all-cause mortality)
Proportion of complications related to the intervention | 90 days after hospital admission
  complications(i.e. major bleeding,minor bleeding, thrombocytopenia) related to the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Zhenguo Zhai, Doctor, Principal Investigator — China-Japan Friendship Hospital
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Piazza G, Rosenbaum EJ, Pendergast W, Jacobson JO, Pendleton RC, McLaren GD, Elliott CG, Stevens SM, Patton WF, Dabbagh O, Paterno MD, Catapane E, Li Z, Goldhaber SZ. Physician alerts to prevent symptomatic venous thromboembolism in hospitalized patients. Circulation. 2009 Apr 28;119(16):2196-201. doi: 10.1161/CIRCULATIONAHA.108.841197. Epub 2009 Apr 13. PMID 19364975
- [Background] Pai M, Lloyd NS, Cheng J, Thabane L, Spencer FA, Cook DJ, Haynes RB, Schunemann HJ, Douketis JD. Strategies to enhance venous thromboprophylaxis in hospitalized medical patients (SENTRY): a pilot cluster randomized trial. Implement Sci. 2013 Jan 2;8:1. doi: 10.1186/1748-5908-8-1. PMID 23279972
- [Background] Kucher N, Koo S, Quiroz R, Cooper JM, Paterno MD, Soukonnikov B, Goldhaber SZ. Electronic alerts to prevent venous thromboembolism among hospitalized patients. N Engl J Med. 2005 Mar 10;352(10):969-77. doi: 10.1056/NEJMoa041533. PMID 15758007
- [Background] Writing Group for the CHECKLIST-ICU Investigators and the Brazilian Research in Intensive Care Network (BRICNet); Cavalcanti AB, Bozza FA, Machado FR, Salluh JI, Campagnucci VP, Vendramim P, Guimaraes HP, Normilio-Silva K, Damiani LP, Romano E, Carrara F, Lubarino Diniz de Souza J, Silva AR, Ramos GV, Teixeira C, Brandao da Silva N, Chang CC, Angus DC, Berwanger O. Effect of a Quality Improvement Intervention With Daily Round Checklists, Goal Setting, and Clinician Prompting on Mortality of Critically Ill Patients: A Randomized Clinical Trial. JAMA. 2016 Apr 12;315(14):1480-90. doi: 10.1001/jama.2016.3463. PMID 27115264
- [Background] Garcia DA, Highfill J, Finnerty K, Varoz E, McConkey S, Hutchinson K, Libby E. A prospective, controlled trial of a pharmacy-driven alert system to increase thromboprophylaxis rates in medical inpatients. Blood Coagul Fibrinolysis. 2009 Oct;20(7):541-5. doi: 10.1097/MBC.0b013e32832d6cfc. PMID 19584716
- [Background] Fontaine A, Mahe I, Bergmann JF, Fiessinger JN, Dhote R, Cohen P, Vinceneux P. Effectiveness of written guidelines on the appropriateness of thromboprophylaxis prescriptions for medical patients: a prospective randomized study. J Intern Med. 2006 Oct;260(4):369-76. doi: 10.1111/j.1365-2796.2006.01699.x. PMID 16961674
- [Derived] Dong F, Zhen K, Zhang Z, Si C, Xia J, Zhang T, Xia L, Wang W, Jia C, Shan G, Zhai Z, Wang C; Chinese Prevention Strategy for Venous Thromboembolism (CHIPS-VTE) study group. Effect on thromboprophylaxis among hospitalized patients using a system-wide multifaceted quality improvement intervention: Rationale and design for a multicenter cluster randomized clinical trial in China. Am Heart J. 2020 Jul;225:44-54. doi: 10.1016/j.ahj.2020.04.020. Epub 2020 May 7. PMID 32474204